CLINICAL TRIAL: NCT05484778
Title: Analysis of Balance and Functional Hop Tests in Athletes With Lower Extremity Injuries by Dual Task Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Aysen Elif Yılmaz, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IU-ELIF-001
Record Dates: First submitted 2022-07-04; First posted 2022-08-02 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Athletic Injuries; Knee Injuries; Ankle Injuries; Hip Injuries; Ankle Sprains; Reinjuries
Keywords: dual-task paradigm
MeSH Terms: conditions — Athletic Injuries; Knee Injuries; Ankle Injuries; Hip Injuries; Reinjuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Group (Other): This group consists of athletes whose are between the ages of 14-30 and are still active at high school or university level in sports involving sudden changes of direction and jump physically and who have a history of injury to only one lower extremity before.
  Interventions: Procedure: Dual tasking paradigm
- Control Group (Other): This group consists of athletes whose age range is 14-30, and who are still active at high school or university level in sports involving sudden changes of direction and jump physically and who do not have a history of lower extremity injuries.
  Interventions: Procedure: Dual tasking paradigm

INTERVENTIONS:
Procedure: Dual tasking paradigm — The dual task methodology is a testing model that requires one person to perform two tasks at the same time. The dual task is divided into two as motor-motor or motor-cognitive. Dual tasks provide an opportunity to examine the attention demands of both tasks and allow possible interference to be observed. The idea behind this design is that central processing capacity has a limit and must be distributed among concurrent tasks.

SUMMARY:
Functional Hop tests and balance measurements are frequently used to decide on returning to sports after lower extremity injuries. Although the athletes show proficiency in these tests and measurements, re-injuries occur when returning to sports. The causes of these re-injuries are mostly functional deficiencies such as inadequate neuromuscular control and stability.

In the competition or sports environment, especially in team games, the athlete also shows cognitive performance, such as communication with teammates and following the game, which are included in the game setup, as well as the physical performance. Performing many tasks or performances at the same time divides the focus of attention on the activities performed, and if the person cannot adequately meet the attention demands, the quality of one or more of the tasks performed will deteriorate. As the level of expertise in the sport increases, the athlete tends to manage his posture, balance and movement with automatic postural control and can focus his attention on a new task.

The concept of focus of attention has been evaluated from different perspectives over time. If it is examined in terms of direction; It is divided into two as the internal focus of attention, which is used by focusing on body movements during the performance of the person, and the external focus of attention, which is used by focusing on the effect of the movement during the performance of the person. As the investigators planned in this study, a second cognitive task assigned to the participant simultaneously during his or her physical performance acts as an external focus of attention, allowing movement control during performance to be carried out by unconscious or automatic processes.

The investigators's aim; It is to examine the balance and functional hop tests that the investigator will apply in athletes by combining them with a simultaneous dual cognitive task that will reflect the field conditions more realistically. In the meantime, investigators think that with the sharing of our results with the literature, it can contribute to both the decision-making processes to return to sports after injury and preventive rehabilitation programs.

DETAILED DESCRIPTION:
As a result of this study, the possible changes in balance and functional jump performances of athletes who have previously had unilateral lower extremity injuries will be examined with the dual-task paradigm. In line with these results, it will be possible to comment on the balance and functional hop test performances of the athletes together with the cognitive task. Balance measurements and functional performance evaluations are used in the decision to return to sports after previous injuries. After the measurements, the affected and unaffected side are compared and an evaluation is made. However, even with these tests and evaluations, athletes are injured again when they return to sports. One of the reasons for this may be that the protective and controlled environment applied during rehabilitation is less challenging and requires less attention when compared to the competitive and sports environment in which the person is involved. For this reason, the investigator think that the evaluations and tests used in the decision to return to sports include both cognitive and physical performance by forcing the attention demands of the person, and it may be more effective in determining the real performance of the person. Thus, the use of physical assessments applied with simultaneous cognitive tasks can be used in the evaluation of the athletes during the return to sports by calculating the possible measurement differences between the affected and unaffected sides compared to the classical procedure, and in the planning of preventive rehabilitation programs of the athletes if there is a decrease in performance in the measurements applied as a dual task. It also contributes to studies that examine performance together with the dual task previously applied to athletes. Secondly, by examining the relationship between balance and functional hop test parameters, it will be determined how effective the independent variables are on each other. If the performance of individuals who have had a previous injury change with the dual task and the mechanisms of these possible changes are known, protective and performance-enhancing strategies can be developed, the cognitive and physical preparation of the athletes for the sports environment can be accelerated, and the risks of re-injury of the athletes can be reduced, as a result of which medical costs can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Having a history of injury to only one lower extremity before
* Having to stay away from sports activities for at least 1 week and maximum 6 weeks after the injury.
* Not having a lower extremity injury in the last 6 months
* Age range of 14-30 and still being active at high school or university level in sports involving sudden changes of direction and jumping physically

Exclusion Criteria:

* Bilateral lower extremity injury history
* Pregnancy
* Vestibular, respiratory and visual disturbances
* Diabetes
* Auditory or cognitive deficit
* Use of drugs that affect balance, cognition and attention
* Pain in the affected lower extremity (at least 2/10 according to the VAS -Visual Analogue Scale-)
* Lower extremity or waist operation history
* Conditions or neurological disorders that may affect balance
* Head trauma or symptoms related to head trauma

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants in the study completed the measurements
Period: Overall Study
Arm/Group | Case Group | Control Group
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Athletes who are still active in team sports (basketball, volleyball and football) that involve sudden changes of direction and jump physically were included in our study. 19 athletes with a history of unilateral lower extremity injuries were divided into the Previously Injured group , and 20 athletes with no previous injury were divided into the Non Injured Group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Case Group | Control Group | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.05 (3.719) | 16.95 (1.395) | 17.97 (2.557)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 1 | 11
  Male | 9 | 19 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Mini Mental State Score [Mean (Standard Deviation); unit: units on a scale] — As a result of the evaluation, a score in the range of 0-30 is obtained. High scores indicate successful and good mental status, while low scores indicate poor results.
  units on a scale | 28.84 (0.688) | 29.35 (0.745) | 29.10 (0.754)
Difficulty Level of Cognitive Task [Mean (Standard Deviation); unit: digits] — This determination method was used in order to personalize the difficulty of the mental task to be used in physical measurements. Each athlete was told a 2-digit random number before the measurements and the athlete was asked to say the same number in reverse. For each correct answer, the number of digits is increased by one. Whichever number of households the participant made a mistake, one more was used in the measurements. And this number of digits was recorded as the cognitive task difficulty level.
  digits | 6.53 (1.020) | 6.30 (0.801) | 6.41 (0.910)
Weight [Mean (Standard Deviation); unit: kilogram] | 69.642 (2.963) | 69.625 (1.284) | 69.633 (9.774)
Height [Mean (Standard Deviation); unit: meter] | 1.804 (0.204) | 1.755 (0.137) | 1.779 (0.079)

OUTCOME MEASURES:

1. Primary Outcome: Balance Performance Measurement (OSI-injured/Worse Side-Single Task)
Description: For balance measurement, Athlete Single Leg Stability, one of the test modes in the Biodex Balance System SD balance device, was preferred. The participant took a position with her/his eyes open, the foot of the untested leg resting on the back of the ankle of the tested leg, her arms crossed over her chest, and the balance center in the middle of the platform most comfortably. The analysis protocol was applied at 5 level, consisting of 20 seconds, 1 sample and 3 test repetitions, with a 10-second rest between repetitions. General stability index (OSI), anterior/posterior stability index (APSI), medial/lateral stability index (MLSI) were recorded.
  The unit of data obtained in this device is the balance index. And values close to 0 indicate high stability.
Time Frame: day 1
Population: Athletes who are still active in team sports (basketball, volleyball and football) that involve sudden changes of direction and jumping were included in our study. 19 athletes with a history of unilateral lower extremity injuries were divided into the Previously Injured group, and 20 athletes with no previous injury were divided into the Non Injured Group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 1.684 (1.034) | 2.300 (0.912)

2. Primary Outcome: Balance Performance Measurement (APSI-injured/Worse Side-Single Task)
Description: as for outcome 1
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 1.131 (0.840) | 1.566 (0.634)

3. Primary Outcome: Balance Performance Measurement (MLSI-injured/Worse Side-Single Task)
Description: as for outcome 1
Time Frame: day 1
Population: Athletes who are still active in team sports (basketball, volleyball and football) that involve sudden changes of direction and jumping were included in our study. 19 athletes with a history of unilateral lower extremity injuries were divided into the Previously Injured group (PIG), and 20 athletes with no previous injury were divided into the Non Injured Group (NIG).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 1.073 (0.565) | 1.405 (0.579)

4. Primary Outcome: Balance Performance Measurement (OSI-noninjured/Better Side-Single Task)
Description: as for outcome 1
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 1.631 (0.958) | 2.725 (1.419)

5. Primary Outcome: Balance Performance Measurement (APSI-noninjured/Better Side- Single Task)
Description: as for outcome 1
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 1.163 (0.621) | 1.770 (0.682)

6. Primary Outcome: Balance Measurement Performance (MLSI-noninjured/Better Side-Single Task)
Description: as for outcome 1
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 0.984 (0.666) | 1.760 (1.392)

7. Primary Outcome: Functional Hop Test (THD-injured/Worse Side-Single Task)
Description: Triple hop for distance ,Crossover hop for distance-CHD -In these two tests, the distance between the starting line and the heel line in step 3 was measured. Normalization was done by dividing this distance (m) by the athlete's height (m).
  The results of this measurement method have certain cut-off values depending on gender and age. In this study, the performance was not compared according to the cut-off values, but between the groups.
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
meter/meter | 2.533 (0.427) | 2.938 (0.441)

8. Primary Outcome: Functional Hop Test (CHD-injured/Worse Side-Single Task)
Description: as for outcome 7
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
meter/meter | 2.366 (0.478) | 2.795 (0.517)

9. Primary Outcome: Functional Hop Test (6MHT-injured/Worse Side-Single Task)
Description: 6m hop for timed-6MTH: The participant was asked to jump on one leg as fast as possible from the marked start point to the finish point, which is 6 meters away from the marked start point. The time from the start to the end of 6 meters was recorded.
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
second | 2.641 (0.337) | 2.374 (0.316)

10. Primary Outcome: Functional Hop Test(THD-noninjured/Better Side- Single Task)
Description: Triple hop for distance ,Crossover hop for distance-CHD -In these two tests, the distance between the starting line and the heel line in step 3 was measured. Normalization was done by dividing this distance (m) by the athlete's height (m).
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
meter/meter | 2.561 (0.447) | 2.950 (0.458)

11. Primary Outcome: Functional Hop Test(CHD-noninjured/Better Side-Single Task)
Description: as for outcome 10
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
meter/meter | 2.350 (0.528) | 2.757 (0.441)

12. Primary Outcome: Functional Hop Test(6MHT-noninjured/Better Side-Single Task)
Description: as for outcome 9
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
second | 2.643 (0.366) | 2.379 (0.371)

13. Primary Outcome: Functional Hop Test THD LSI-Single Task
Description: The limb symmetry index (LSI) was calculated to evaluate the difference between the two legs in all functional tests. Calculation for the case group; LSI = Affected leg score ÷ Unaffected leg score × 100 This calculation for the control group; LSI= Worse score ÷ Better score × 100.
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of leg's performance
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
percentage of leg's performance | 99.586 (9.879) | 95.643 (5.387)

14. Primary Outcome: Functional Hop Test CHD LSI-Single Task
Description: as for outcome 13
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of leg's performance
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
percentage of leg's performance | 101.627 (10.415) | 91.766 (5.650)

15. Primary Outcome: Functional Hop Test 6MHT LSI-Single Task
Description: as for outcome 13
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of leg's performance
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
percentage of leg's performance | 100.181 (7.505) | 92.794 (8.541)

16. Secondary Outcome: Balance Performance Measurement (OSI-injured/Worse Side-Dual Task)
Description: as for outcome 1
Time Frame: day 1
Population: Athletes who are still active in team sports (basketball, volleyball and football) that involve sudden changes of direction and jumping were included in our study. 19 athletes with a history of unilateral lower extremity injuries were divided into the Previously Injured group, and 20 athletes with no previous injury were divided into the Non Injured Group .
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 1.652 (0.826) | 2.138 (0.903)

17. Secondary Outcome: Balance Performance Measurement (APSI-injured/Worse Side-Dual Task)
Description: as for outcome 1
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 1.078 (0.646) | 1.377 (0.627)

18. Secondary Outcome: Balance Performance Measurement (MLSI-injured/Worse Side-Dual Task)
Description: as for outcome 1
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 1.073 (0.508) | 1.400 (0.773)

19. Secondary Outcome: Balance Performance Measurement (OSI-noninjured/Better Side- Dual Task)
Description: as for outcome 1
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 1.605 (0.687) | 2.555 (1.648)

20. Secondary Outcome: Balance Performance Measurement(APSI-noninjured/Better Side-Dual Task)
Description: as for outcome 1
Time Frame: day 1
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 1.142 (0.567) | 1.475 (0.517)

21. Secondary Outcome: Balance Performance Measurement(MLSI-noninjured/Better Side-Dual Task)
Description: as for outcome 1
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
score on a scale | 0.952 (0.400) | 1.805 (1.696)

22. Secondary Outcome: Functional Hop Test(THD-injured/Worse Side-Dual Task)
Description: as for outcome 10
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
meter/meter | 2.531 (0.436) | 2.908 (0.473)

23. Secondary Outcome: Functional Hop Test (CHD-injured/Worse Side-Dual Task)
Description: as for outcome 10
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
meter/meter | 2.362 (0.431) | 2.774 (0.467)

24. Secondary Outcome: Functional Hop Test (6MHT-injured/Worse Side-Dual Task)
Description: as for outcome 9
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
second | 2.732 (0.404) | 2.496 (0.459)

25. Secondary Outcome: Functional Hop Test(THD-noninjured/Better Side-Dual Task)
Description: as for outcome 10
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
meter/meter | 2.543 (0.449) | 2.966 (0.481)

26. Secondary Outcome: Functional Hop Test(CHD-noninjured/Better Side-Dual Task)
Description: as for outcome 10
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
meter/meter | 2.406 (0.488) | 2.773 (0.461)

27. Secondary Outcome: Functional Hop Test(6MHT-noninjured/Better Side-Dual Task)
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
second | 2.755 (0.404) | 2.462 (0.378)

28. Secondary Outcome: Functional Hop Test THD LSI-Dual Task
Description: as for outcome 13
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of leg's performance
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
percentage of leg's performance | 100.042 (8.549) | 95.666 (4.276)

29. Secondary Outcome: Functional Hop Test CHD LSI-Dual Task
Description: as for outcome 13
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of leg's performance
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
percentage of leg's performance | 98.888 (10.218) | 94.587 (4.513)

30. Secondary Outcome: Functional Hop Test 6MHT LSI-Dual Task
Description: as for outcome 13
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of leg's performance
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 19 | 20
percentage of leg's performance | 101.154 (7.694) | 93.315 (4.265)

ADVERSE EVENTS:
Time Frame: Adverse event data not collected
Description: The tests used in the study are the RTS (return the sport) tests applied to the athletes. There is no risk of adverse effects as these tests are performed in the clinic and under supervision.
Arm/Group | Case Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT05484778/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT05484778/SAP_001.pdf